CLINICAL TRIAL: NCT01705938
Title: A First In Human, Single Blind, Placebo Controlled, Randomized Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SP-333 Tablets in Healthy Adult Subjects
Brief Title: Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of SP-333 Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: SP333101
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Exposure
MeSH Terms: interventions — dolcanatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Group 1 (Active Comparator): SP-333 0.1 mg & Placebo, one tablet by mouth, single dose
  Interventions: Drug: SP-333
- Group 2 (Active Comparator): SP-333 0.3 mg & Placebo, 3 tablets by mouth, single dose
  Interventions: Drug: SP-333
- Group 3 (Active Comparator): SP-333 1 mg & Placebo, one tablet by mouth, single dose
  Interventions: Drug: SP-333
- Group 4 (Active Comparator): SP-333 3 mg & Placebo, 3 tablets by mouth,single dose
  Interventions: Drug: SP-333
- Group 5 (Active Comparator): SP-333 10 mg & Placebo, 1 tablet by mouth, single dose
  Interventions: Drug: SP-333
- Group 6 (Active Comparator): SP-333 30 mg & Placebo, 3 tablets by mouth, single dose
  Interventions: Drug: SP-333
- Group 7 (Active Comparator): SP-333 60 mg & Placebo, 6 tablets by mouth, single dose
  Interventions: Drug: SP-333

INTERVENTIONS:
Drug: SP-333

SUMMARY:
This is a randomized, phase 1, single-blind, placebo-controlled, randomized, sequential, escalating, single-dose, study designed to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) properties of orally administered SP-333 tablets.

DETAILED DESCRIPTION:
This is a randomized, phase 1, single-blind, placebo controlled, single-dose, study designed to evaluate the safety, tolerability, and pharmacokinetic properties of orally administered SP-333 tablets. The study will include 7 groups of 8 subjects each (6 active, 2 placebo) given a single oral dose of of SP-333 tablets or placebo. Following outpatient screening from approximately 5 to 42 days before dosing, each subject will enter the Clinical Pharmacology Unit (CPU) and will be housed from at least 48 hours, before dosing until 48 hours after dosing. Subjects will be given single dose of the study drug on the day of dosing and remain in the CPU for at least 48 hours. Subjects will return to the CPU on Days 8±1 and 15±1 for safety follow up. Safety Committee Meetings will be conducted to review safety, tolerability, and available Pharmacokinetic data from the current and previous treatment group(s), prior to dosing subsequent treatment groups. Subjects in a given treatment group are considered completers once they have completed the Day 15±1 day Follow up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 55 years old
2. Body weight greater than or equal to 50 kg (110 pounds) and Body Mass Index (BMI) in the range of 18 to 30 kg/ m2
3. Medically healthy with no clinically significant findings.
4. Subjects must have bowel habits that are considered regular (for this study a minimum of 4 bowel movements a week without laxatives).
5. Subject must have had a bowel movement, without laxatives, in the 3 days before administration of study drug.
6. Male subjects with female sexual partners of child-bearing potential must agree to use highly effective contraceptive methods during the study.
7. Female subjects must be post-menopausal and not pregnant.
8. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign an Informed Consent Form.

Exclusion Criteria:

1. Smokers or users of nicotine products who do not agree to not smoke or use nicotine products during their stay in the CPU.
2. Current or history of clinically significant diseases, including gastrointestinal, renal, hepatic, neurologic (e.g., neuropathy), hematologic, endocrine (e.g., diabetes), oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition.
3. Presence of any abnormal clinically significant laboratory.
4. History of any serious allergic reaction to any medication
5. Certain abnormalities of the ECG.
6. Participated in a previous clinical study with an investigational product within 30 days of study Participation
7. Donated blood, blood components or significant loss of blood within 2 months of dosing
8. History of a clinically-significant illness within 4 weeks of dosing
9. Special diet, any dietary habits, or restrictions, which, may interfere with conduct of the study or health of the subject within 30 days of dosing
10. History of clinically-significant drug or alcohol abuse within 2 years of study participation
11. Positive urine screen for prohibited drugs (cocaine, cannabinoids, opiates, barbiturates, amphetamines, benzodiazepines, phencyclidine, propoxyphene).
12. History of human immunodeficiency virus (HIV), hepatitis B surface antigen positive (+HBsAg), or hepatitis C antibody positive (+HCVAb).
13. History of certain surgeries:

    * Gastric bypass surgery or invasive procedure for the treatment of obesity or surgery to remove a segment of the gastrointestinal (GI) tract at any time.
    * Patients who have had a gastric band (unless the band has been completely removed for more than 60 days)
    * Surgery of the abdomen, pelvis or retroperitoneal structures within six months of study participation.
    * Appendectomy,Instrumentation of the bowel, major surgery within 60 days of study participation.
14. Female subjects of childbearing potential or who are breastfeeding
15. Use of any routine systemic medication, including any over the counter (OTC) medication within 2 weeks of dosing
16. Use of herbal products, dietary supplements, vitamins, grapefruit, or grapefruit containing products within 2 weeks of dosing
17. Irregular daily bowel habits
18. Any other issue which, in the judgment of the investigator, will make the subject ineligible for study participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with treatment emergent adverse events as a measure of safety and tolerability | 14 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of SP-333 following single oral doses of tablets. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Peter Winkle, MD, Principal Investigator — Anaheim Clinical Trials
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States